CLINICAL TRIAL: NCT02557399
Title: Clinical Evaluation of Efficacy at 2 Weeks of Duac® Fixed Dose Combination Gel in Treatment of Facial Acne Vulgaris in Japanese Subjects
Brief Title: DUAC® Early Onset Efficacy Study in Japanese Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201884
Record Dates: First submitted 2015-06-11; First posted 2015-09-23 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris
Keywords: Clindamycin; Gel; Benzoyl Peroxide; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination; Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duac® fixed dose combination gel (Experimental): Subjects will use Duac® fixed dose combination gel (clindamycin phosphate 1.2% and benzoyl peroxide 3%) with quantity sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) for 12 weeks.
  Interventions: Drug: Duac® fixed dose combination gel
- Combination therapy: ADA 0.1% gel + CLDM 1% gel (Active Comparator): Subjects will use combination therapy of ADA 0.1% gel with quantity sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) and subjects will also apply CLDM 1% gel twice daily, once in the morning and once in the evening (at bedtime) for 12 weeks. The CLDM 1% gel should apply subsequent to the application of ADA 0.1% gel in the evening. The CLDM 1% gel should be applied to ILs only.
  Interventions: Drug: ADA 0.1% gel; Drug: CLDM 1% gel

INTERVENTIONS:
Drug: Duac® fixed dose combination gel — Duac® fixed dose combination gel containing clindamycin phosphate 1.2% and benzoyl peroxide 3%.
  Arms: Duac® fixed dose combination gel
Drug: ADA 0.1% gel — ADA 0.1% gel containing 0.1% of adapalene.
  Arms: Combination therapy: ADA 0.1% gel + CLDM 1% gel
Drug: CLDM 1% gel — CLDM 1% gel containing clindamycin phosphate 1.2% (1% as clindamycin).
  Arms: Combination therapy: ADA 0.1% gel + CLDM 1% gel

SUMMARY:
This is a multicentre, randomized, single-blind (investigator is blinded), active (the combination therapy of adapalene [ADA] and clindamycin [CLDM])-controlled and parallel-group study in Japanese subjects with facial acne vulgaris. The purpose of this study is to evaluate the efficacy, safety and tolerability of CLDM 1 percent (%)-benzoyl peroxide 3% (Duac®: trademark owned by GlaxoSmithKline) once daily fixed dose combination gel versus combination therapy of ADA 0.1% gel and CLDM 1% gel in the topical treatment of facial acne vulgaris for 12 weeks. A total of 400 subjects will be screened for enrolment. Subjects will use Duac® fixed dose combination gel with quantity sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) or combination therapy of ADA 0.1% gel with quantity sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) and CLDM 1% gel twice daily, once in the morning and once in the evening (at bedtime) for 12 weeks.

DETAILED DESCRIPTION:
Duac® is a registered trademark of Stiefel Laboratories, Inc., a GSK company. Duac® marketed in Japan is CLDM 1%-benzoyl peroxide 3% combination gel.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 12 to 45 years of age, inclusive.
* Subjects must have had both: (a) A minimum of 17 but not more than 60 ILs (papules / pustules) on the face, including nasal lesions; (b) A minimum of 20 but not more than 150 non-ILs (open / closed comedones) on the face, including nasal lesions.
* Subjects who have an ISGA score of 2 or greater at Baseline.
* Female subjects of childbearing potential and women who are less than 2 years from their last menses must agree to use contraception
* Subjects who are willing and able to follow all study procedures and to visit all scheduled evaluation points.
* Subjects who have ability to understand and give a written informed consent form (written informed consent must be obtained also from the parent or guardian if the participant is under 20 years of age).

Exclusion Criteria:

* Subjects who have any nodulo-cystic lesions at Baseline.
* Female subjects who are pregnant or who are breast-feeding.
* Subjects who have a history or presence of regional enteritis, inflammatory bowel disease (e.g. ulcerative colitis, pseudomembranous colitis, chronic diarrhoea, antibiotic-associated colitis or bloody diarrhoea) or similar symptoms.
* Subjects who used any of the following agents within 2 weeks prior to Baseline: topical antibiotics on the face or systemic antibiotics; topical anti-acne medications (e.g. Benzoyl peroxide, azelaic acid, resorcinol, salicylates etc.); abradants, facials, peels, masks containing glycolic or other acids; washes, soaps, non mild facial cleansers containing benzoyl peroxide, salicylic acid or sulfacetamide sodium; moisturizers containing retinol, salicylic acid or alpha or beta-hydroxy acids (except additive agent); astringents and toner.
* Subjects who used any of the following agents on the face or performed the following procedure within 4 weeks prior to baseline: topical corticosteroids applied onto face (use of inhaled, intra-articular or intra-lesional steroids other than for facial acne is acceptable); facial procedure (such as chemical and laser peel, microdermabration, blue light treatment, etc.).
* Subjects who used systemic retinoids within the previous 6 months or topical retinoids within 6 weeks prior to Baseline.
* Subjects who received treatment with estrogens, androgens or anti-androgenic agents within the previous 12 weeks (subjects who have been treated with the above agents for more than 12 consecutive weeks prior to start of investigational product are allowed to enrol as long as they do not expect to change dose, drug or discontinue use during the study).
* Subjects who are using any medication that in the opinion of the investigator may affect this clinical study or evaluation of the study.
* Subjects who plan to use medications that are reported to exacerbate acne (such as vitamin D and vitamin B12, corticosteroids, androgens, haloperidol, halogens, lithium, hydantoin and Phenobarbital).
* Subjects who have a known hypersensitivity or have had previous allergic reaction to any of the components of the investigational product.
* Subjects who have used investigate therapy within the previous 12 weeks or plan to participate in another clinical study at the same time.
* Subjects who participated in another Japanese clinical study planned by GlaxoSmithKline K.K. in the development of investigational products for acne vulgaris.
* Subjects with a history of substance abuse (alcohol or drugs) or substance dependence within 12 months prior to screening.
* Subjects who have medical history suggestive of an immunocompromized status.
* Subjects who are employees of a GlaxoSmithKline, an investigator or clinical research organization involved in the study or any immediate family member of an employee involved in the study.
* Subjects who have any other condition that would put the subject at unacceptable risk for participation in the study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2016-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Japan (6):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: DUAC® (clindamycin phosphate 1.2 percent [%] + benzoyl peroxide 3%) is the registered product of GlaxoSmithKline. This study was conducted between 07 October 2015 and 17 February 2016 in which 349 participants were randomized.
Groups:
- DUAC: Participants were instructed to use DUAC, a fixed dose combination gel (clindamycin phosphate 1.2% and benzoyl peroxide 3%) with quantity of 2 finger tip unit (FTU) about 0.6 gram (g) which was sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) for 12 weeks.
- ADA 0.1% +CLDM 1%: Participants were instructed to use combination therapy of Adapalene (ADA) 0.1% gel with quantity of 1 FTU about 0.5 g sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) and clindamycin (CLDM) 1% gel twice daily, once in the morning and once in the evening (at bedtime) for 12 weeks. The CLDM 1% gel was applied subsequent to the application of ADA 0.1% gel in the evening. The CLDM 1% gel was applied to inflammatory lesions (ILs) only.
Period: Overall Study
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Started | 172 | 177
Completed | 165 | 169
Not Completed | 7 | 8
Not completed — Adverse Event | 6 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Protocol-defined stopping criteria | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- DUAC: Participants were instructed to use DUAC, a fixed dose combination gel (clindamycin phosphate 1.2% and benzoyl peroxide 3%) with quantity equal to about 0.6 g which was sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) for 12 weeks.
- ADA 0.1% +CLDM 1%: Participants were instructed to use combination therapy of ADA 0.1% gel with quantity equal to about 0.5 g sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) and CLDM 1% gel twice daily, once in the morning and once in the evening (at bedtime) for 12 weeks. The CLDM 1% gel was applied subsequent to the application of ADA 0.1% gel in the evening. The CLDM 1% gel was applied to ILs only.
- Total: Total of all reporting groups
Arm/Group | DUAC | ADA 0.1% +CLDM 1% | Total
Number analyzed (Participants) | 172 | 177 | 349
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.3 (5.91) | 19.8 (4.90) | 20.0 (5.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 110 | 207
  Male | 75 | 67 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 172 | 177 | 349
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Lesion Counts (TLs) From Baseline to Week 2
Description: The assessor performed a count of IL (papules, pustules, nodular lesions), non-ILs (open and closed comedones) and total lesions (the sum of IL and non-IL) at each study visit. Lesion counts were confined to the face. Change from Baseline was calculated as the value at endpoint minus the value at Baseline. Data for adjusted mean has been reported. Percent change from Baseline is the change from Baseline divided by Baseline value multiplied by 100. The Baseline value was the latest pre-dose assessment value. The non-inflammatory lesions were counted by diagnosis based on palpation of the investigator (or sub-investigator).
Time Frame: Baseline (Day 1) and Week 2
Population: Intent-to-Treat (ITT) population comprised of all randomized participants who received at least one application of study product. Only those participants with data available at the indicated time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Percent change in lesions
Groups:
- DUAC: Participants were instructed to use DUAC, a fixed dose combination gel (clindamycin phosphate 1.2% and benzoyl peroxide 3%) with quantity of 2 FTU about 0.6 gram (g) which was sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) for 12 weeks.
- ADA 0.1% +CLDM 1%: Participants were instructed to use combination therapy of ADA 0.1% gel with quantity of 1 FTU about 0.5 g sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) and CLDM 1% gel twice daily, once in the morning and once in the evening (at bedtime) for 12 weeks. The CLDM 1% gel was applied subsequent to the application of ADA 0.1% gel in the evening. The CLDM 1% gel was applied to ILs only.
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 169 | 176
Percent change in lesions | -42.16 (1.890) | -35.33 (1.850)
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.008, mixed model repeated measures analysis — The analysis method was mixed model repeated measures analysis with treatment, center, visit, treatment-by-visit interaction, Baseline TLs counts, Baseline-by-visit interaction as fixed effects; difference in percent = -6.83, 95% CI 2-sided [-11.88 to -1.78] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM

2. Secondary Outcome: Percent Change From Baseline in TLs to Weeks 1, 4, 8 and 12
Description: The assessor performed a count of IL (papules, pustules, nodular lesions), non-ILs (open and closed comedones) and total lesions (the sum of IL and non-IL) at each study visit. Lesion counts were confined to the face. Change from Baseline was calculated as the value at endpoint minus the value at Baseline. Data for adjusted mean has been reported. Percent change from Baseline is the change from Baseline divided by Baseline value multiplied by 100. The Baseline value was the latest pre-dose assessment value. The non-ILs were counted by diagnosis based on palpation of the investigator (or sub-investigator). A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM.
Time Frame: Baseline (Day 1) and Week 1, 4, 8, 12
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change in lesions
Groups:
- DUAC: Participants were instructed to use DUAC, a fixed dose combination gel (clindamycin phosphate 1.2% and benzoyl peroxide 3%) with quantity of 2 FTU about 0.6 g which was sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) for 12 weeks.
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Percent change in lesions
  Week 1: number analyzed (Participants) | 172 | 176
  Week 1 | -24.58 (1.729) | -24.33 (1.697)
  Week 4: number analyzed (Participants) | 169 | 174
  Week 4 | -55.51 (1.670) | -49.65 (1.637)
  Week 8: number analyzed (Participants) | 167 | 172
  Week 8 | -65.23 (1.544) | -62.88 (1.514)
  Week 12: number analyzed (Participants) | 164 | 169
  Week 12 | -74.60 (1.314) | -71.36 (1.288)
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.916, mixed model repeated measures analysis — The analysis method was mixed-model for repeated measures with treatment, center, visit, treatment-by-visit interaction, Baseline TLs counts, Baseline-by-visit interaction as fixed effects; difference in percent = -0.25, 95% CI 2-sided [-4.85 to 4.35] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1
Statistical Analysis 2: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.010, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; difference in percent = -5.85, 95% CI 2-sided [-10.29 to -1.42] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4
Statistical Analysis 3: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.257, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; difference in percent = -2.35, 95% CI 2-sided [-6.42 to 1.72] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8
Statistical Analysis 4: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.062, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; difference in percent = -3.24, 95% CI 2-sided [-6.64 to 0.16] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12

3. Secondary Outcome: Percent Change Form Baseline in Lesion Counts (ILs and Non-ILs) to Weeks 1, 2, 4, 8 and 12
Description: The assessor performed a count of IL (papules, pustules, nodular lesions), non-ILs (open and closed comedones). Lesion counts were confined to the face. Change from Baseline was calculated as the value at endpoint minus the value at Baseline. Data for adjusted mean has been reported. Percent change from Baseline is the change from Baseline divided by Baseline value multiplied by 100. The Baseline value was the latest pre-dose assessment value. The non-ILs were counted by diagnosis based on palpation of the investigator (or sub-investigator).
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, 12
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change in lesions
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Percent change in lesions
  Week 1 ILs: number analyzed (Participants) | 172 | 176
  Week 1 ILs | -42.97 (2.349) | -37.89 (2.309)
  Week 2 ILs: number analyzed (Participants) | 169 | 176
  Week 2 ILs | -60.92 (2.209) | -52.49 (2.162)
  Week 4 ILs: number analyzed (Participants) | 169 | 174
  Week 4 ILs | -70.68 (1.898) | -61.30 (1.860)
  Week 8 ILs: number analyzed (Participants) | 167 | 172
  Week 8 ILs | -76.33 (1.717) | -69.64 (1.682)
  Week 12 ILs: number analyzed (Participants) | 164 | 169
  Week 12 ILs | -82.07 (1.403) | -77.58 (1.374)
  Week 1 non-ILs: number analyzed (Participants) | 172 | 176
  Week 1 non-ILs | -15.13 (2.279) | -17.85 (2.239)
  Week 2 non-ILs: number analyzed (Participants) | 169 | 176
  Week 2 non-ILs | -32.71 (2.419) | -27.01 (2.367)
  Week 4 non-ILs: number analyzed (Participants) | 169 | 174
  Week 4 non-ILs | -47.64 (2.171) | -43.74 (2.129)
  Week 8 non-ILs: number analyzed (Participants) | 167 | 172
  Week 8 non-ILs | -59.50 (1.910) | -58.91 (1.872)
  Week 12 non-ILs: number analyzed (Participants) | 164 | 169
  Week 12 non-ILs | -71.07 (1.603) | -67.29 (1.571)
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.115, mixed model repeated measures analysis — The analysis method was mixed-model for repeated measures with treatment, center, visit, treatment-by-visit interaction, Baseline ILs counts, Baseline-by-visit interaction as fixed effects; difference in percent = -5.08, 95% CI 2-sided [-11.41 to 1.25] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1 for ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 2: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.005, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; difference in percent = -8.43, 95% CI 2-sided [-14.35 to -2.51] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2 for ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 3: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p < 0.001, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; difference in percent = -9.37, 95% CI 2-sided [-14.42 to -4.33] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4 for ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 4: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.004, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; difference in percent = -6.69, 95% CI 2-sided [-11.21 to -2.16] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8 for ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 5: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.015, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -4.50, 95% CI 2-sided [-8.10 to -0.89] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12 for ILs
Statistical Analysis 6: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.382, mixed model repeated measures analysis — The analysis method was mixed-model for repeated measures with treatment, center, visit, treatment-by-visit interaction, Baseline non-ILs counts, Baseline-by-visit interaction as fixed effects; difference in percent = 2.71, 95% CI 2-sided [-3.38 to 8.80] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1 for non-ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 7: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.085, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; difference in percent = -5.69, 95% CI 2-sided [-12.17 to 0.78] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2 for non-ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 8: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.186, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; difference in percent = -3.89, 95% CI 2-sided [-9.67 to 1.88] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4 for non-ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 9: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.818, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; difference in percent = -0.59, 95% CI 2-sided [-5.61 to 4.44] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8 for non-ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 10: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.073, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; difference in percent = -3.78, 95% CI 2-sided [-7.92 to 0.35] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12 for non-ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM

4. Secondary Outcome: Absolute Change From Baseline in Lesion Counts (TLs, ILs and Non-ILs) to Weeks 1, 2, 4, 8 and 12
Description: The assessor performed a count of IL (papules, pustules, nodular lesions), non-ILs (open and closed comedones) and total lesions (the sum of IL and non-IL) at each study visit. Lesion counts were confined to the face. Change from Baseline was calculated as the value at endpoint minus the value at Baseline. Data for adjusted mean has been reported. The non-ILs were counted by diagnosis based on palpation of the investigator (or sub-investigator). A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM. The Baseline value was the latest pre-dose assessment value.
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, 12
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
lesion count
  Week 1 TLs: number analyzed (Participants) | 172 | 176
  Week 1 TLs | -24.4 (1.70) | -24.3 (1.67)
  Week 2 TLs: number analyzed (Participants) | 169 | 176
  Week 2 TLs | -41.8 (1.88) | -35.6 (1.84)
  Week 4 TLs: number analyzed (Participants) | 169 | 174
  Week 4 TLs | -56.3 (1.71) | -51.6 (1.67)
  Week 8 TLs: number analyzed (Participants) | 167 | 172
  Week 8 TLs | -66.4 (1.60) | -65.7 (1.57)
  Week 12 TLs: number analyzed (Participants) | 164 | 169
  Week 12 TLs | -76.2 (1.37) | -74.5 (1.34)
  Week 1 ILs: number analyzed (Participants) | 172 | 176
  Week 1 ILs | -13.3 (0.74) | -11.5 (0.72)
  Week 2 ILs: number analyzed (Participants) | 169 | 176
  Week 2 ILs | -19.3 (0.70) | -16.3 (0.68)
  Week 4 ILs: number analyzed (Participants) | 169 | 174
  Week 4 ILs | -22.4 (0.62) | -19.8 (0.60)
  Week 8 ILs: number analyzed (Participants) | 167 | 172
  Week 8 ILs | -24.3 (0.56) | -22.4 (0.55)
  Week 12 ILs: number analyzed (Participants) | 164 | 169
  Week 12 ILs | -26.0 (0.48) | -24.9 (0.47)
  Week 1 non-ILs: number analyzed (Participants) | 172 | 176
  Week 1 non-ILs | -11.1 (1.46) | -12.9 (1.43)
  Week 2 non-ILs: number analyzed (Participants) | 169 | 176
  Week 2 non-ILs | -22.5 (1.59) | -19.3 (1.56)
  Week 4 non-ILs: number analyzed (Participants) | 169 | 174
  Week 4 non-ILs | -34.0 (1.46) | -32.0 (1.44)
  Week 8 non-ILs: number analyzed (Participants) | 167 | 172
  Week 8 non-ILs | -42.2 (1.33) | -43.4 (1.31)
  Week 12 non-ILs: number analyzed (Participants) | 164 | 169
  Week 12 non-ILs | -50.2 (1.11) | -49.6 (1.09)
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.961, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.1, 95% CI 2-sided [-4.6 to 4.4] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1 for TLs. negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 2: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.015, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -6.2, 95% CI 2-sided [-11.2 to -1.2] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2 for TLs. negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 3: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.044, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -4.7, 95% CI 2-sided [-9.2 to -0.1] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4 for TLs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 4: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.747, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-4.9 to 3.5] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8 for TLs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 5: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.338, mixed model repeated measures analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.7, 95% CI 2-sided [-5.3 to 1.8] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12 for TLs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 6: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.068, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.8 to 0.1] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.002, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -3.0, 95% CI 2-sided [-4.8 to -1.1] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.002, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -2.6, 95% CI 2-sided [-4.3 to -1.0] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 9: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.012, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -1.9, 95% CI 2-sided [-3.4 to -0.4] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 10: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.078, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.4 to 0.1] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12 for ILs. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 11: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.367, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; Mean Difference (Net) = 1.8, 95% CI 2-sided [-2.1 to 5.7] — [estimate comment as in outcome 3, analysis 6]
Statistical Analysis 12: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.148, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; Mean Difference (Net) = -3.1, 95% CI 2-sided [-7.4 to 1.1] — [estimate comment as in outcome 3, analysis 7]
Statistical Analysis 13: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.314, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; Mean Difference (Net) = -2.0, 95% CI 2-sided [-5.9 to 1.9] — [estimate comment as in outcome 3, analysis 8]
Statistical Analysis 14: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.494, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; Mean Difference (Net) = 1.2, 95% CI 2-sided [-2.3 to 4.7] — [estimate comment as in outcome 3, analysis 9]
Statistical Analysis 15: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.684, mixed model repeated measures analysis — [p-value comment as in outcome 3, analysis 6]; Mean Difference (Net) = -0.6, 95% CI 2-sided [-3.5 to 2.3] — [estimate comment as in outcome 3, analysis 10]

5. Secondary Outcome: Percentage of Participants With a Minimum of 2-grade Improvement in Investigator's Static Global Assessment (ISGA) Score From Baseline to Weeks 1, 2, 4, 8 and 12
Description: Responder was defined as participants with a minimum 2-grade improvement in ISGA score from Baseline. ISGA scale was scored from 0-5 (0= Clear skin with no inflammatory or non-ILs, 1= Almost clear: rare non-ILs present, with no more than rare papules, 2= Mild severity: greater than Grade 1, some non-ILs with no more than few inflammatory lesions, 3= Moderate severity: greater than Grade 2, many non-ILS, may have some ILs, but no more than 1 small nodular lesion, 4= Severe: greater than Grade 3, up to many non-ILs and ILs, but no more than a few nodular lesions, 5= Very severe: many non -ILs and ILs and more than a few nodular lesions. May have cystic lesions). Percentage of participants was calculated by dividing number of participants with 2-grade improvement in ISGA score from Baseline by total number of participants value multiplied by 100.
Time Frame: Week 1, 2, 4, 8, 12
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Percentage of participants
  Week 1 | 2 | 0
  Week 2 | 6 | 3
  Week 4 | 12 | 8
  Week 8 | 22 | 12
  Week 12 | 37 | 27
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 2.3, 95% CI 2-sided [0.1 to 4.6] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1.The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 2: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.185, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 3.0, 95% CI 2-sided [-1.3 to 7.3] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 3: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.251, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 3.7, 95% CI 2-sided [-2.5 to 9.9] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 4: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 10.2, 95% CI 2-sided [2.4 to 18.0] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 5: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 10.7, 95% CI 2-sided [0.9 to 20.4] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit

6. Secondary Outcome: Percentage of Participants With ISGA Score of 0 or 1 at Weeks 1, 2, 4, 8 and 12
Description: Responder was defined as participant with ISGA score of 0 or 1. ISGA scale was scored from 0-5 (0= Clear skin with no inflammatory or non-ILs, 1= Almost clear: rare non-ILs present, with no more than rare papules, 2= Mild severity: greater than Grade 1, some non-ILs with no more than few inflammatory lesions, 3= Moderate severity: greater than Grade 2, many non-ILS, may have some ILs, but no more than 1 small nodular lesion, 4= Severe: greater than Grade 3, up to many non-ILs and ILs, but no more than a few nodular lesions, 5= Very severe: many non -ILs and ILs and more than a few nodular lesions. May have cystic lesions). Percentage of participants was calculated by dividing number of participants with 0-1 ISGA score post Baseline by total number of participants value multiplied by 100.
Time Frame: Week 1, 2, 4, 8 and 12
Population: ITT population.
Measure: Number; unit: Percentage of participants
Groups:
- ADA 0.1% +CLDM 1%: Participants were instructed to use combination therapy of ADA) 0.1% gel with quantity of 1 FTU about 0.5 g sufficient to cover entire face (including the forehead, nose, cheeks and chin) once daily in the evening (at bedtime) and CLDM 1% gel twice daily, once in the morning and once in the evening (at bedtime) for 12 weeks. The CLDM 1% gel was applied subsequent to the application of ADA 0.1% gel in the evening. The CLDM 1% gel was applied to ILs only.
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Percentage of participants
  Week 1 | 2 | 1
  Week 2 | 6 | 5
  Week 4 | 13 | 6
  Week 8 | 20 | 12
  Week 12 | 41 | 29
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.129, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 1.8, 95% CI 2-sided [-0.7 to 4.3] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 2: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.612, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 1.3, 95% CI 2-sided [-3.4 to 5.9] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 7.1, 95% CI 2-sided [1.1 to 13.2] — [estimate comment as in outcome 5, analysis 3]
Statistical Analysis 4: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 7.9, 95% CI 2-sided [0.3 to 15.5] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 5: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 11.3, 95% CI 2-sided [1.4 to 21.3] — [estimate comment as in outcome 5, analysis 5]

7. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in Lesion Counts (TLs, ILs and Non-ILs) From Baseline at Weeks 1, 2, 4, 8 and 12
Description: Responder was defined as participants with at least a 50% reduction in TLs, ILs and non-ILs. Data for number of participants is reported. Percentage of participants was calculated by dividing number of responders by total number of participants value multiplied by 100.
Time Frame: Week 1, 2, 4, 8 and 12
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Percentage of participants
  Week 1 TLs: number analyzed (Participants) | 172 | 176
  Week 1 TLs | 22 | 18
  Week 2 TLs | 47 | 42
  Week 4 TLs | 67 | 60
  Week 8 TLs | 81 | 81
  Week 12 TLs | 88 | 86
  Week 1 ILs: number analyzed (Participants) | 172 | 176
  Week 1 ILs | 51 | 42
  Week 2 ILs | 77 | 66
  Week 4 ILs | 85 | 76
  Week 8 ILs | 87 | 84
  Week 12 ILs | 92 | 89
  Week 1 non-ILs: number analyzed (Participants) | 172 | 176
  Week 1 non-ILs | 14 | 16
  Week 2 non-ILs | 37 | 34
  Week 4 non-ILs | 58 | 54
  Week 8 non-ILs | 73 | 73
  Week 12 non-ILs | 83 | 80
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.379, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 3.9, 95% CI 2-sided [-4.5 to 12.3] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1 for TLs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 2: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.409, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 4.7, 95% CI 2-sided [-5.7 to 15.1] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2 for TLs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 3: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.180, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 7.0, 95% CI 2-sided [-3.1 to 17.0] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4 for TLs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 4: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.810, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = -0.5, 95% CI 2-sided [-8.8 to 7.7] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8 for TLs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 5: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.648, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 1.9, 95% CI 2-sided [-5.2 to 9.0] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12 for TLs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 6: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 9.1, 95% CI 2-sided [-1.3 to 19.6] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1 for ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 7: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 11.2, 95% CI 2-sided [1.8 to 20.6] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2 for ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 8: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.044, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 8.6, 95% CI 2-sided [0.4 to 16.9] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4 for ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 9: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.345, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 3.6, 95% CI 2-sided [-3.8 to 11.0] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8 for ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 10: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.424, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 2.6, 95% CI 2-sided [-3.5 to 8.7] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12 for ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 11: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.527, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = -2.0, 95% CI 2-sided [-9.4 to 5.5] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 1 for non-ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 12: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.584, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 3.3, 95% CI 2-sided [-6.7 to 13.4] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 2 for non-ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 13: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.519, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = 3.9, 95% CI 2-sided [-6.5 to 14.3] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4 for non-ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 14: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.766, Cochran-Mantel-Haenszel — The P-values are based on the Cochran-Mantel-Haenszel test stratified by center; Difference in percentage = -0.8, 95% CI 2-sided [-10.1 to 8.5] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8 for non-ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit
Statistical Analysis 15: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.666, Cochran-Mantel-Haenszel — The P-value was based on the Cochran-Mantel-Haenszel test stratified by center; Odds Ratio (OR) = 2.3, 95% CI 2-sided [-5.8 to 10.5] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12 for non-ILs. The participants with missing data at a visit were included in the denominator (n) at the visit. That is, those participants were treated as non-responder at the visit

8. Secondary Outcome: Number of Participants With Treatment Adherence Rate at Weeks 1, 2, 4, 8 and 12
Description: The investigator (or sub-investigator), the product storage manager, or the blinded coordinator dispensed a study compliance log to record participant's compliance with investigational product application from Baseline to the end of study treatment. The product storage manager or the blinded coordinator evaluated the participant's compliance with study treatment, using the study compliance log at each visit, and recorded the compliance data in the eCRF.
Time Frame: Week 1, 2, 4, 8 and 12
Population: ITT population.
Measure: Number; unit: Participants
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Participants
  week 1 | 143 | 131
  week 2 | 125 | 115
  week 4 | 110 | 85
  week 8 | 89 | 72
  week 12 | 88 | 63

9. Secondary Outcome: Number of Participants Who Continued Treatment at Weeks 1, 2, 4, 8 and 12
Description: Number of participants who continued the treatment till Week 12 was measured. Overall data for participants who have not missed any dose during the treatment period has been reported.
Time Frame: Up to Week 12
Population: ITT population.
Measure: Number; unit: Participants
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Participants | 63 | 59

10. Secondary Outcome: Participant's Treatment Preference at Weeks 1, 2, 4, 8 and 12
Description: Participants had to rate each question on a 5-point scale of 0 to 4 (4: yes, very easy to use, 3: yes, easy, 2: slightly easy, 1: slightly difficult, 0: No) where larger score indicates more preferable participant's feeling. There were 5 questions in the questionnaire: ease of application, comfort, satisfaction with treatment (ST), comparison with prior therapies (CPT) and willingness to continue using the product (WCP).
Time Frame: Week 1, 2, 4, 8 and 12
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Participants
  Week 1: Ease of application, Score 4: number analyzed (Participants) | 172 | 176
  Week 1: Ease of application, Score 4 | 131 | 95
  Week 1: Ease of application, Score 3: number analyzed (Participants) | 172 | 176
  Week 1: Ease of application, Score 3 | 38 | 66
  Week 1: Ease of application, Score 2: number analyzed (Participants) | 172 | 176
  Week 1: Ease of application, Score 2 | 2 | 13
  Week 1: Ease of application, Score 1: number analyzed (Participants) | 172 | 176
  Week 1: Ease of application, Score 1 | 1 | 2
  Week 2: Ease of application, Score 4: number analyzed (Participants) | 169 | 176
  Week 2: Ease of application, Score 4 | 128 | 83
  Week 2: Ease of application, Score 3: number analyzed (Participants) | 169 | 176
  Week 2: Ease of application, Score 3 | 38 | 75
  Week 2: Ease of application, Score 2: number analyzed (Participants) | 169 | 176
  Week 2: Ease of application, Score 2 | 2 | 17
  Week 2: Ease of application, Score 1: number analyzed (Participants) | 169 | 176
  Week 2: Ease of application, Score 1 | 1 | 1
  Week 4: Ease of application, Score 4: number analyzed (Participants) | 169 | 174
  Week 4: Ease of application, Score 4 | 118 | 85
  Week 4: Ease of application, Score 3: number analyzed (Participants) | 169 | 174
  Week 4: Ease of application, Score 3 | 49 | 70
  Week 4: Ease of application, Score 2: number analyzed (Participants) | 169 | 174
  Week 4: Ease of application, Score 2 | 2 | 18
  Week 4: Ease of application, Score 1: number analyzed (Participants) | 169 | 174
  Week 4: Ease of application, Score 1 | 0 | 1
  Week 8: Ease of application, Score 4: number analyzed (Participants) | 167 | 172
  Week 8: Ease of application, Score 4 | 114 | 90
  Week 8: Ease of application, Score 3: number analyzed (Participants) | 167 | 172
  Week 8: Ease of application, Score 3 | 50 | 60
  Week 8: Ease of application, Score 2: number analyzed (Participants) | 167 | 172
  Week 8: Ease of application, Score 2 | 3 | 19
  Week 8: Ease of application, Score 1: number analyzed (Participants) | 167 | 172
  Week 8: Ease of application, Score 1 | 0 | 3
  Week 12: Ease of application, Score 4: number analyzed (Participants) | 164 | 169
  Week 12: Ease of application, Score 4 | 116 | 81
  Week 12: Ease of application, Score 3: number analyzed (Participants) | 164 | 169
  Week 12: Ease of application, Score 3 | 44 | 68
  Week 12: Ease of application, Score 2: number analyzed (Participants) | 164 | 169
  Week 12: Ease of application, Score 2 | 4 | 18
  Week 12: Ease of application, Score 1: number analyzed (Participants) | 164 | 169
  Week 12: Ease of application, Score 1 | 0 | 2
  Week 1: Comfort, Score 4: number analyzed (Participants) | 172 | 176
  Week 1: Comfort, Score 4 | 37 | 24
  Week 1: Comfort, Score 3: number analyzed (Participants) | 172 | 176
  Week 1: Comfort, Score 3 | 86 | 69
  Week 1: Comfort, Score 2: number analyzed (Participants) | 172 | 176
  Week 1: Comfort, Score 2 | 37 | 45
  Week 1: Comfort, Score 1: number analyzed (Participants) | 172 | 176
  Week 1: Comfort, Score 1 | 7 | 32
  Week 1: Comfort, Score 0: number analyzed (Participants) | 172 | 176
  Week 1: Comfort, Score 0 | 5 | 6
  Week 2: Comfort, Score 4: number analyzed (Participants) | 169 | 176
  Week 2: Comfort, Score 4 | 56 | 35
  Week 2: Comfort, Score 3: number analyzed (Participants) | 169 | 176
  Week 2: Comfort, Score 3 | 70 | 81
  Week 2: Comfort, Score 2: number analyzed (Participants) | 169 | 176
  Week 2: Comfort, Score 2 | 36 | 42
  Week 2: Comfort, Score 1: number analyzed (Participants) | 169 | 176
  Week 2: Comfort, Score 1 | 6 | 17
  Week 2: Comfort, Score 0: number analyzed (Participants) | 169 | 176
  Week 2: Comfort, Score 0 | 1 | 1
  Week 4: Comfort, Score 4: number analyzed (Participants) | 169 | 174
  Week 4: Comfort, Score 4 | 72 | 47
  Week 4: Comfort, Score 3: number analyzed (Participants) | 169 | 174
  Week 4: Comfort, Score 3 | 75 | 80
  Week 4: Comfort, Score 2: number analyzed (Participants) | 169 | 174
  Week 4: Comfort, Score 2 | 17 | 31
  Week 4: Comfort, Score 1: number analyzed (Participants) | 169 | 174
  Week 4: Comfort, Score 1 | 5 | 15
  Week 4: Comfort, Score 0: number analyzed (Participants) | 169 | 174
  Week 4: Comfort, Score 0 | 0 | 1
  Week 8: Comfort, Score 4: number analyzed (Participants) | 167 | 172
  Week 8: Comfort, Score 4 | 79 | 53
  Week 8: Comfort, Score 3: number analyzed (Participants) | 167 | 172
  Week 8: Comfort, Score 3 | 69 | 68
  Week 8: Comfort, Score 2: number analyzed (Participants) | 167 | 172
  Week 8: Comfort, Score 2 | 18 | 36
  Week 8: Comfort, Score 1: number analyzed (Participants) | 167 | 172
  Week 8: Comfort, Score 1 | 1 | 13
  Week 8: Comfort, Score 0: number analyzed (Participants) | 167 | 172
  Week 8: Comfort, Score 0 | 0 | 2
  Week 12: Comfort, Score 4: number analyzed (Participants) | 164 | 169
  Week 12: Comfort, Score 4 | 84 | 56
  Week 12: Comfort, Score 3: number analyzed (Participants) | 164 | 169
  Week 12: Comfort, Score 3 | 66 | 73
  Week 12: Comfort, Score 2: number analyzed (Participants) | 164 | 169
  Week 12: Comfort, Score 2 | 13 | 26
  Week 12: Comfort, Score 1: number analyzed (Participants) | 164 | 169
  Week 12: Comfort, Score 1 | 1 | 13
  Week 12: Comfort, Score 0: number analyzed (Participants) | 164 | 169
  Week 12: Comfort, Score 0 | 0 | 1
  Week 1: ST, Score 4: number analyzed (Participants) | 172 | 176
  Week 1: ST, Score 4 | 36 | 21
  Week 1: ST, Score 3: number analyzed (Participants) | 172 | 176
  Week 1: ST, Score 3 | 79 | 75
  Week 1: ST, Score 2: number analyzed (Participants) | 172 | 176
  Week 1: ST, Score 2 | 46 | 49
  Week 1: ST, Score 1: number analyzed (Participants) | 172 | 176
  Week 1: ST, Score 1 | 11 | 23
  Week 1: ST, Score 0: number analyzed (Participants) | 172 | 176
  Week 1: ST, Score 0 | 0 | 8
  Week 2: ST, Score 4: number analyzed (Participants) | 169 | 176
  Week 2: ST, Score 4 | 58 | 38
  Week 2: ST, Score 3: number analyzed (Participants) | 169 | 176
  Week 2: ST, Score 3 | 70 | 81
  Week 2: ST, Score 2: number analyzed (Participants) | 169 | 176
  Week 2: ST, Score 2 | 37 | 47
  Week 2: ST, Score 1: number analyzed (Participants) | 169 | 176
  Week 2: ST, Score 1 | 4 | 7
  Week 2: ST, Score 0: number analyzed (Participants) | 169 | 176
  Week 2: ST, Score 0 | 0 | 3
  Week 4: ST, Score 4: number analyzed (Participants) | 169 | 174
  Week 4: ST, Score 4 | 66 | 44
  Week 4: ST, Score 3: number analyzed (Participants) | 169 | 174
  Week 4: ST, Score 3 | 72 | 81
  Week 4: ST, Score 2: number analyzed (Participants) | 169 | 174
  Week 4: ST, Score 2 | 27 | 40
  Week 4: ST, Score 1: number analyzed (Participants) | 169 | 174
  Week 4: ST, Score 1 | 4 | 8
  Week 4: ST, Score 0: number analyzed (Participants) | 169 | 174
  Week 4: ST, Score 0 | 0 | 1
  Week 8: ST, Score 4: number analyzed (Participants) | 167 | 172
  Week 8: ST, Score 4 | 78 | 58
  Week 8: ST, Score 3: number analyzed (Participants) | 167 | 172
  Week 8: ST, Score 3 | 67 | 72
  Week 8: ST, Score 2: number analyzed (Participants) | 167 | 172
  Week 8: ST, Score 2 | 17 | 33
  Week 8: ST, Score 1: number analyzed (Participants) | 167 | 172
  Week 8: ST, Score 1 | 5 | 6
  Week 8: ST, Score 0: number analyzed (Participants) | 167 | 172
  Week 8: ST, Score 0 | 0 | 3
  Week 12: ST, Score 4: number analyzed (Participants) | 164 | 169
  Week 12: ST, Score 4 | 82 | 63
  Week 12: ST, Score 3: number analyzed (Participants) | 164 | 169
  Week 12: ST, Score 3 | 61 | 70
  Week 12: ST, Score 2: number analyzed (Participants) | 164 | 169
  Week 12: ST, Score 2 | 20 | 29
  Week 12: ST, Score 1: number analyzed (Participants) | 164 | 169
  Week 12: ST, Score 1 | 1 | 6
  Week 12: ST, Score 0: number analyzed (Participants) | 164 | 169
  Week 12: ST, Score 0 | 0 | 1
  Week 1: CPT, Score 4: number analyzed (Participants) | 172 | 176
  Week 1: CPT, Score 4 | 77 | 53
  Week 1: CPT, Score 3: number analyzed (Participants) | 172 | 176
  Week 1: CPT, Score 3 | 50 | 45
  Week 1: CPT, Score 2: number analyzed (Participants) | 172 | 176
  Week 1: CPT, Score 2 | 38 | 61
  Week 1: CPT, Score 1: number analyzed (Participants) | 172 | 176
  Week 1: CPT, Score 1 | 7 | 11
  Week 1: CPT, Score 0: number analyzed (Participants) | 172 | 176
  Week 1: CPT, Score 0 | 0 | 6
  Week 2: CPT, Score 4,: number analyzed (Participants) | 169 | 176
  Week 2: CPT, Score 4, | 90 | 57
  Week 2: CPT, Score 3: number analyzed (Participants) | 169 | 176
  Week 2: CPT, Score 3 | 51 | 55
  Week 2: CPT, Score 2: number analyzed (Participants) | 169 | 176
  Week 2: CPT, Score 2 | 25 | 54
  Week 2: CPT, Score 1: number analyzed (Participants) | 169 | 176
  Week 2: CPT, Score 1 | 2 | 10
  Week 2: CPT, Score 0: number analyzed (Participants) | 169 | 176
  Week 2: CPT, Score 0 | 1 | 0
  Week 4: CPT, Score 4: number analyzed (Participants) | 169 | 174
  Week 4: CPT, Score 4 | 100 | 67
  Week 4: CPT, Score 3: number analyzed (Participants) | 169 | 174
  Week 4: CPT, Score 3 | 47 | 52
  Week 4: CPT, Score 2: number analyzed (Participants) | 169 | 174
  Week 4: CPT, Score 2 | 18 | 46
  Week 4: CPT, Score 1: number analyzed (Participants) | 169 | 174
  Week 4: CPT, Score 1 | 4 | 8
  Week 4: CPT, Score 0: number analyzed (Participants) | 169 | 174
  Week 4: CPT, Score 0 | 0 | 1
  Week 8: CPT, Score 4: number analyzed (Participants) | 167 | 172
  Week 8: CPT, Score 4 | 109 | 73
  Week 8: CPT, Score 3: number analyzed (Participants) | 167 | 172
  Week 8: CPT, Score 3 | 38 | 50
  Week 8: CPT, Score 2: number analyzed (Participants) | 167 | 172
  Week 8: CPT, Score 2 | 19 | 40
  Week 8: CPT, Score 1: number analyzed (Participants) | 167 | 172
  Week 8: CPT, Score 1 | 1 | 8
  Week 8: CPT, Score 0: number analyzed (Participants) | 167 | 172
  Week 8: CPT, Score 0 | 0 | 1
  Week 12: CPT, Score 4: number analyzed (Participants) | 164 | 169
  Week 12: CPT, Score 4 | 112 | 78
  Week 12: CPT, Score 3: number analyzed (Participants) | 164 | 169
  Week 12: CPT, Score 3 | 42 | 47
  Week 12: CPT, Score 2: number analyzed (Participants) | 164 | 169
  Week 12: CPT, Score 2 | 8 | 35
  Week 12: CPT, Score 1: number analyzed (Participants) | 164 | 169
  Week 12: CPT, Score 1 | 2 | 7
  Week 12: CPT, Score 0: number analyzed (Participants) | 164 | 169
  Week 12: CPT, Score 0 | 0 | 2
  Week 1: WCP, Score 4: number analyzed (Participants) | 172 | 176
  Week 1: WCP, Score 4 | 64 | 36
  Week 1: WCP, Score 3: number analyzed (Participants) | 172 | 176
  Week 1: WCP, Score 3 | 79 | 78
  Week 1: WCP, Score 2: number analyzed (Participants) | 172 | 176
  Week 1: WCP, Score 2 | 25 | 39
  Week 1: WCP, Score 1: number analyzed (Participants) | 172 | 176
  Week 1: WCP, Score 1 | 4 | 19
  Week 1: WCP, Score 0: number analyzed (Participants) | 172 | 176
  Week 1: WCP, Score 0 | 0 | 4
  Week 2: WCP, Score 4: number analyzed (Participants) | 169 | 176
  Week 2: WCP, Score 4 | 75 | 55
  Week 2: WCP, Score 3: number analyzed (Participants) | 169 | 176
  Week 2: WCP, Score 3 | 72 | 70
  Week 2: WCP, Score 2: number analyzed (Participants) | 169 | 176
  Week 2: WCP, Score 2 | 19 | 38
  Week 2: WCP, Score 1: number analyzed (Participants) | 169 | 176
  Week 2: WCP, Score 1 | 3 | 13
  Week 4: WCP, Score 4: number analyzed (Participants) | 169 | 174
  Week 4: WCP, Score 4 | 88 | 63
  Week 4: WCP, Score 3: number analyzed (Participants) | 169 | 174
  Week 4: WCP, Score 3 | 63 | 75
  Week 4: WCP, Score 2: number analyzed (Participants) | 169 | 174
  Week 4: WCP, Score 2 | 15 | 26
  Week 4: WCP, Score 1: number analyzed (Participants) | 169 | 174
  Week 4: WCP, Score 1 | 3 | 10
  Week 8: WCP, Score 4: number analyzed (Participants) | 167 | 172
  Week 8: WCP, Score 4 | 90 | 62
  Week 8: WCP, Score 3: number analyzed (Participants) | 167 | 172
  Week 8: WCP, Score 3 | 59 | 74
  Week 8: WCP, Score 2: number analyzed (Participants) | 167 | 172
  Week 8: WCP, Score 2 | 15 | 27
  Week 8: WCP, Score 1: number analyzed (Participants) | 167 | 172
  Week 8: WCP, Score 1 | 3 | 9
  Week 12: WCP, Score 4: number analyzed (Participants) | 164 | 169
  Week 12: WCP, Score 4 | 94 | 70
  Week 12: WCP, Score 3: number analyzed (Participants) | 164 | 169
  Week 12: WCP, Score 3 | 56 | 65
  Week 12: WCP, Score 2: number analyzed (Participants) | 164 | 169
  Week 12: WCP, Score 2 | 12 | 23
  Week 12: WCP, Score 1: number analyzed (Participants) | 164 | 169
  Week 12: WCP, Score 1 | 1 | 11
  Week 12: WCP, Score 0: number analyzed (Participants) | 164 | 169
  Week 12: WCP, Score 0 | 1 | 0

11. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Score at Week 2, 4, 8 and 12
Description: QOL questionnaire was assessed using Skindex-16 with 16 questions in 3 multi-item scales: symptoms, emotions and functioning for the past week: skin condition-itching, burning or stinging, hurting, being irritated, persistence/reoccurrence of skin condition, worry about condition, appearance of skin, frustration about skin, embarrassment about skin, being annoyed about your skin, feeling depressed about skin, effects of your skin on your interactions with others, effects of your skin condition on your desire to be with people, skin condition making it hard to show affection, effects of your skin condition on your daily activities and skin condition making it hard to work or do what you enjoy. Data for adjusted mean has been reported. The Baseline value was the latest pre-dose assessment value. Change from Baseline was calculated as the value at endpoint minus the value at Baseline. Scores range from 0-never bothered to 100-always bothered.
Time Frame: Baseline(Day 1) and Week 2, 4, 8 and 12
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Score on scale
  Week 2: number analyzed (Participants) | 169 | 176
  Week 2 | -0.71 (0.070) | -0.49 (0.068)
  Week 4: number analyzed (Participants) | 169 | 174
  Week 4 | -1.02 (0.069) | -0.80 (0.068)
  Week 8: number analyzed (Participants) | 167 | 172
  Week 8 | -1.14 (0.073) | -0.92 (0.071)
  Week 12: number analyzed (Participants) | 164 | 169
  Week 12 | -1.27 (0.073) | -1.10 (0.072)
Statistical Analysis 1: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.017, mixed model repeated measures analysis; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.40 to -0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.017, mixed model repeated measures analysis; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.40 to -0.04] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 4. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 3: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.024, mixed model repeated measures analysis; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.41 to -0.03] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 8. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM
Statistical Analysis 4: Comparison: DUAC vs ADA 0.1% +CLDM 1%; Test type: Superiority or Other; p = 0.080, mixed model repeated measures analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.36 to 0.02] — Comparison between DUAC and ADA 0.1% +CLDM 1% at Week 12. A negative treatment difference indicates a benefit of Duac relative to ADA+CLDM

12. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Medical or scientific judgment was exercised in deciding whether reporting was appropriate. For liver injury and impaired liver function, alanine aminotransferase greater than or equal to (>=)3 times upper limit of normal (ULN) and total bilirubin >=2xULN (less than [>] 35% direct) was defined.
Time Frame: Up to Week 12
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Participants
  Any AE | 53 | 100
  Any SAE | 1 | 0

13. Secondary Outcome: Local Tolerability Score for Erythema, Dryness, Peeling, Itching, and Burning or Stinging
Description: Local tolerability score for erythema (no redness, faint red or pink coloration, barely perceptible, light red or pink coloration, medium red coloration, beet red coloration), dryness (none, barely perceptible dryness with no flakes or fissure formation, easily perceptible dryness with no flakes or fissure formation, easily noted dryness and flakes but no fissure formation, easily noted dryness with flakes and fissure formation), peeling (no peeling, mild localized peeling, mild and diffuse peeling, moderate and diffuse peeling, moderate to prominent, dense peeling) and itching and burning/stinging (normal-no discomfort, noticeable discomfort that causes intermittent awareness, continuous awareness, intermittent awareness and interferes occasionally with normal daily activities, a definite continuous discomfort that interferes with normal daily activities) was assessed on a scale of 0 to 4 (0= absent, 1= slight, 2= mild, 3= moderate and 4= severe).
Time Frame: Week 1, 2, 4, 8 and 12
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Score on scale
  Erythema Week 1: number analyzed (Participants) | 170 | 175
  Erythema Week 1 | 0.0 (0.61) | 0.3 (0.72)
  Erythema Week 2: number analyzed (Participants) | 169 | 175
  Erythema Week 2 | 0.0 (0.68) | 0.0 (0.70)
  Erythema Week 4: number analyzed (Participants) | 169 | 174
  Erythema Week 4 | -0.1 (0.57) | -0.1 (0.64)
  Erythema Week 8: number analyzed (Participants) | 165 | 171
  Erythema Week 8 | -0.2 (0.68) | -0.2 (0.69)
  Erythema Week 12: number analyzed (Participants) | 165 | 168
  Erythema Week 12 | -0.2 (0.78) | -0.3 (0.67)
  Dryness Week 1: number analyzed (Participants) | 170 | 175
  Dryness Week 1 | 0.1 (0.54) | 0.6 (0.95)
  Dryness Week 2: number analyzed (Participants) | 169 | 175
  Dryness Week 2 | 0.0 (0.50) | 0.1 (0.58)
  Dryness Week 4: number analyzed (Participants) | 169 | 174
  Dryness Week 4 | 0.0 (0.52) | 0.1 (0.49)
  Dryness Week 8: number analyzed (Participants) | 165 | 171
  Dryness Week 8 | 0.0 (0.58) | 0.1 (0.46)
  Dryness Week 12: number analyzed (Participants) | 165 | 168
  Dryness Week 12 | 0.0 (0.45) | 0.0 (0.35)
  Peeling Week 1: number analyzed (Participants) | 170 | 175
  Peeling Week 1 | 0.1 (0.43) | 0.5 (0.88)
  Peeling Week 2: number analyzed (Participants) | 169 | 175
  Peeling Week 2 | 0.1 (0.33) | 0.2 (0.55)
  Peeling Week 4: number analyzed (Participants) | 169 | 174
  Peeling Week 4 | 0.0 (0.34) | 0.1 (0.42)
  Peeling Week 8: number analyzed (Participants) | 165 | 171
  Peeling Week 8 | 0.1 (0.39) | 0.1 (0.46)
  Peeling Week 12: number analyzed (Participants) | 165 | 168
  Peeling Week 12 | 0.0 (0.31) | 0.0 (0.32)
  Itching Week 1: number analyzed (Participants) | 170 | 175
  Itching Week 1 | 0.0 (0.64) | 0.1 (0.81)
  Itching Week 2: number analyzed (Participants) | 169 | 175
  Itching Week 2 | 0.0 (0.60) | 0.1 (0.77)
  Itching Week 4: number analyzed (Participants) | 169 | 174
  Itching Week 4 | -0.1 (0.68) | -0.1 (0.62)
  Itching Week 8: number analyzed (Participants) | 165 | 171
  Itching Week 8 | -0.2 (0.63) | -0.1 (0.58)
  Itching Week 12: number analyzed (Participants) | 165 | 168
  Itching Week 12 | -0.2 (0.66) | -0.2 (0.56)
  Burning/Stinging Week 1: number analyzed (Participants) | 170 | 175
  Burning/Stinging Week 1 | 0.0 (0.48) | 0.5 (0.85)
  Burning/Stinging Week 2: number analyzed (Participants) | 169 | 175
  Burning/Stinging Week 2 | 0.0 (0.44) | 0.2 (0.66)
  Burning/Stinging Week 4: number analyzed (Participants) | 169 | 174
  Burning/Stinging Week 4 | 0.0 (0.44) | 0.0 (0.47)
  Burning/Stinging Week 8: number analyzed (Participants) | 165 | 171
  Burning/Stinging Week 8 | 0.0 (0.34) | 0.1 (0.53)
  Burning/Stinging Week 12: number analyzed (Participants) | 165 | 168
  Burning/Stinging Week 12 | 0.0 (0.39) | 0.0 (0.40)

14. Secondary Outcome: Number of Participants With Severity of AEs
Description: The severity of AEs was assessed by the investigator; events were assigned to one of the following categories: mild, an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; moderate, an event that was sufficiently discomforting to interfere with normal everyday activities; and severe, an event that prevented normal everyday activities.
Time Frame: Up to Week 12
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DUAC | ADA 0.1% +CLDM 1%
Number analyzed (Participants) | 172 | 177
Participants
  Mild | 46 | 91
  Modertae | 6 | 7
  Severe | 1 | 2

ADVERSE EVENTS:
Time Frame: AE and SAE were collected up to Week 12.
Description: For AE and SAE, ITT population was analyzed.
Arm/Group | Duac | ADA 0.1% +CLDM 1%
Serious Adverse Events (participants affected / at risk) | 1/172 | 0/177
Other Adverse Events (participants affected / at risk) | 34/172 | 78/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duac (N=172) | ADA 0.1% +CLDM 1% (N=177)
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duac (N=172) | ADA 0.1% +CLDM 1% (N=177)
Application site dryness (General disorders) | 16 (16) | 44 (46)
Nasopharyngitis (Infections and infestations) | 12 (13) | 15 (16)
Application site pain (General disorders) | 3 (3) | 20 (21)
Application site erythema (General disorders) | 4 (4) | 11 (12)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.